CLINICAL TRIAL: NCT04782882
Title: Effectiveness of Progressive Muscle Relaxation and Laughter Therapy on Mental Health and Treatment Outcomes in Women Undergoing In Vitro Fertilization: A Randomized Controlled Trial
Brief Title: The Effect of Progressive Muscle Relaxation and Laughter Therapy on Women Undergoing In Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Sibel Kıyak, Assist. Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NecmettinEU_Kiyak1
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistical and reporting blinding were provided in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In the first session of the researcher (S.K.), the participants were explained the effects of anxiety and stress on the treatment in simple terms for 5 min. Then, information was given about the effects of laughter therapy and progressive muscle relaxation on the body. Laughter therapy was applied for 15-20 min. Then, the lights were turned off and progressive muscle relaxation exercises were performed for 15-20 min under candlelight and accompanied by music. The procedures were received as a group (2-6 people) in 3-4 face-to-face sessions.
  Interventions: Behavioral: Progressive muscle relaxation+laughter therapy
- Control group (No Intervention): The control group then received routine care

INTERVENTIONS:
Behavioral: Progressive muscle relaxation+laughter therapy — Laughter therapy:Laughter therapy is a technique that changes the mood by breathing correctly and by combining childish exercises with laughter exercises to turn into real laughter for no reason.
  Progressive muscle relaxation procedure:
  the participants were asked to tighten and relax large muscle groups in the body with deep breathing exercises. Progressive muscle relaxation was applied to the muscles of the head and face, neck, chest, back, arms, hands, abdomen, hips, legs and feet. The procedure was applied in a dark environment and accompanied by candlelight and relaxing music.
  Arms: intervention group

SUMMARY:
Purpose: This study was aimed to evaluate the effect of progressive muscle relaxation exercises and laughter therapy on the mental health and treatment outcomes of women receiving IVF treatment.

Design: Randomized controlled trial with two parallel groups Methods: Participants were randomly assigned to the intervention (IG; n = 71) and control group (CG; n = 70). The progressive muscle relaxation and laughter therapy was administered to women in the intervention group in the IVF center for 3-4 times and 40 minutes. The CG received routine care. Data were collected using baseline and oocyte retrieval day STAI and BDI.

DETAILED DESCRIPTION:
Infertility, one of the important components of reproductive health, affects one in four couples in developing countries.The emergence of assisted reproductive techniques such as in vitro fertilization (IVF) gives infertile couples the opportunity to have both pregnancy and a baby. Couples are affected emotionally during IVF treatment and women experience more problems than men. The majority of women experience emotional problems such as anxiety and depression because of infertility, invasive treatment procedures, physiological effects of gonadotropin stimulation and positive outcome expectation.Considering the effect of anxiety and depression on infertile women, it is important to examine the effectiveness of progressive muscle relaxation exercises and laughter therapy as complementary therapy in psychosocial care.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 20 and 46,
* Literate in Turkish language,
* Diagnosed with infertility by an obstetrician or medical doctor
* Those with primary or secondary infertility

Exclusion Criteria:

* A diagnosed psychiatric disorder,
* prior experience in relaxation intervention,
* Lack of ovarian response in previous treatments
* Undergoing frozen embryo transfer.

Ages: 20 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Mental health state (anxiety) | Before intervention begins and through intervention completion on average of 15 days
  Beck Depression Inventory: The Beck Depression Inventory (BDI) is a 21-item self-reporting scale consisting of emotional, cognitive, somatic, and motivational components to measure the level and severity changes of depressive symptoms. In BDI, it is seen that as the total score obtained from the scale increases, the individual's level of experiencing depressive emotions increases proportionally.
Mental health state (Depression) | Before intervention begins and through intervention completion on average of 15 days
  State Trait Anxiety Inventory (STAI): To measure anxiety levels of the participants, the Turkish version of STAI developed by Spielberger was used. High scores indicate high anxiety level, while low scores indicate less anxiety level.

SECONDARY OUTCOMES:
Fertility treatment results | Before intervention begins and a cycle of ovarian stimulation (15 days)
  Estradiol (E2) level
Fertility treatment results | a cycle of ovarian stimulation (15 days)
  oocyte count
Fertility treatment results | 3-5 days after oocyte pick up day
  embryo transfer status
Fertility treatment results | 15 days after embryo transfer
  Rate of positive Hcg blood pregnancy test

CONTACTS AND LOCATIONS:
Locations (1):
- Sibel KİYAK, Selçuklu, Konya, Turkey (Türkiye)